CLINICAL TRIAL: NCT02005445
Title: Obstructive Sleep Apnea Treatment to Improve Cardiac Rehabilitation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to meet recruitment target
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F1351-P
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Obstructive Sleep Apnea; Coronary Heart Disease
Keywords: Obstructive sleep apnea; Coronary heart disease; Cardiac rehabilitation; Cardiopulmonary exercise testing
MeSH Terms: conditions — Sleep Apnea, Obstructive; Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Continuous Positive Airway Pressure (CPAP) (Experimental): Continuous positive airway pressure
  Interventions: Device: CPAP
- Healthy Lifestyle and Sleep Education (HLSE) (Sham Comparator): Healthy living and sleep education
  Interventions: Behavioral: HLSE

INTERVENTIONS:
Device: CPAP — Continuous positive airway pressure
  Arms: Continuous Positive Airway Pressure (CPAP)
Behavioral: HLSE — Healthy living and sleep education
  Arms: Healthy Lifestyle and Sleep Education (HLSE)

SUMMARY:
This is a randomized clinical trial in U.S. Veterans to evaluate the impact of treatment for obstructive sleep apnea (OSA) on the effectiveness of cardiac rehabilitation, including impact on exercise capacity, disability, and quality of life.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a highly prevalent condition in patients with coronary heart disease and is associated with impaired exercise performance, functional limitation and reduced health-related quality of life. The investigators hypothesize that identification and treatment of OSA in patients undergoing cardiac rehabilitation will improve the response to rehabilitation. The proposed study will test this hypothesis using a parallel group, randomized, clinical trial comparing OSA treatment with continuous positive airway pressure (CPAP) to an educational control group in patients undergoing cardiac rehabilitation who screen positive for previously undiagnosed OSA.

ELIGIBILITY:
Inclusion Criteria:

* Veterans referred for cardiac rehabilitation at the VA Boston Healthcare System.
* Moderate to severe OSA (AHI >15) on home sleep testing.

Exclusion Criteria:

* Dangerous levels of sleepiness (Epworth Sleepiness Scale score >16 or a report of falling asleep at the wheel of a car within the past 2 years).
* Physical limitation precluding exercise testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Gottlieb, MD MPH, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CPAP | HLSE
Started | 2 | 2
Completed | 2 | 1
Not Completed | 0 | 1
Not completed — Dual study enrollment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPAP | HLSE | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Apnea-hypopnea index [Median (Full Range); unit: events/hour] — Based on 3% desaturation criterion for hypopneas; measured on a continuous scale in events per hour
  events/hour | 19.7 [19.3 to 20.0] | 25.8 [19.8 to 31.7] | 19.9 [19.3 to 31.7]

OUTCOME MEASURES:

1. Primary Outcome: WHO Disability Assessment Scale 2 Scores
Description: Functional status as measured by the World Health Organization Disability Assessment Scale 2.0. Score range 0-48 (higher scores indicate more disability).
Time Frame: 12 weeks
Population: As we were unable to recruit a sufficient number of patients for meaningful analysis, due to closing of the cardiac Rehabilitation program, no analysis was performed. Because there were only 1-2 participants completing the study in each arm, data are not presented due too confidentiality concerns.
Arm/Group | CPAP | HLSE
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | CPAP | HLSE
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPAP (N=2) | HLSE (N=2)
Chest Pain (Cardiac disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT02005445/Prot_SAP_000.pdf